CLINICAL TRIAL: NCT05704010
Title: Role of Videocapsule Endoscopy in Lynch Syndrome: a Multicenter Italian Registry Study
Brief Title: Videocapsule Endoscopy in Lynch Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Raffaele University (Other)
Collaborators: Unita' di Gastroenterologia - Policlinico Universitario di Bari (Unknown); Unita' di Gastroenterologia - Centro di Riferimento Oncologico di Aviano (Unknown); Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Cavestro Giulia Martina MD PhD, Prof Cavestro Giulia Martina, San Raffaele University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Lynch&VCE/01/2018
Record Dates: First submitted 2023-01-13; First posted 2023-01-30 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Lynch Syndrome; Lynch Syndrome I; Lynch Syndrome II; MLH1 Gene Mutation; MSH2 Gene Mutation; MSH6 Gene Mutation; PMS2 Gene Mutation; Small Bowel Adenocarcinoma
Keywords: Videocapsule; Small bowel
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Lynch Syndrome II | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lynch Syndrome (Experimental): Video capsule endoscopy every 2 years
  Interventions: Device: Video capsule endoscopy

INTERVENTIONS:
Device: Video capsule endoscopy — Video capsule endoscopy every 2 years

SUMMARY:
Background Lynch syndrome is caused by a pathogenic variant in one of the four Mismatch Repair genes (MMR): MLH1, MSH2/Epcam, MSH6, or PMS2. These pathogenic variants confer a higher risk of developing colorectal and other cancers, including small bowel cancer. The risk of developing a small bowel adenocarcinoma is about 100 times higher compared to individuals without Lynch syndrome, and the lifetime risk of small bowel cancer is estimated at 4,2%.

The diagnosis of a small bowel cancer depends on videocapsule endoscopy (VCE). This device is swalled so that it can record images of the small bowel, which are then stored on a wearable device for about 8 hours. The capsule is then expelled in the feces while the images are transferred to a computer to be analysed. To date, there is conflicting evidence on the efficacy of small bowel cancer screening with VCE

Rationale: this registry study will collect prospective data from patients with LS undergoing VCE

Aim: evaluate the incidence of neoplastic and pre-neoplastic lesions in patients with LS during a VCE-based small bowel cancer screening study

Design: this is a multicentric, observational study that analyzes data from diagnostic techniques already approved. Patients will not undergo diagnostic procedures beyond what would be recommended by clinical practice.

DETAILED DESCRIPTION:
Background Lynch syndrome (LS) is caused by a pathogenic germline defect in one of the mismatch repair genes (MMR), namely MLH1, MSH2/Epcam, MSH6, or PMS2. Such pathogenic defects confer a higher risk of developing not only colorectal cancer but also small bowel cancer (SBC). Patients with LS have a lifetime risk of SMB of 4.2%, with a relative risk of >100, compared to the general population. Moreover, patients with LS may develop SBC at a younger age, compared to SBC in individuals without LS.

The diagnostic standard for SBC is video capsule endoscopy (VCE). This consists in swallowing a pill with a camera inside. The VCE will record the images through the gastrointestinal tract and send them via Bluetooth to a wearable device for roughly 8 hours The capsule is then expelled with feces while the images are stored in a computer for later revision. Today, the data on the efficacy of a screening program for SBC in patients with LS is controversial.

Rationale This register study will collect prospective data on the VCEs done on patients with LS

Objective To estimate the incidence of neoplasia and preneoplastic lesions of the small bowel in patients with LS via VCE

Design Multicentric observational study with the use of approved diagnostic devices. It will not modify the current standard of care. The study design will not mandate obligatory studies of further procedures besides those that are clinically approved.

Population At least 10 subjects/year by each center (400 patients by study completion)

Controindications to VCE

* Stenosis, obstructions, fistulas (suspected or known)
* Cardiac defibrillators or cardiac pace-makers.
* Dysphagia
* Inability to provide written informed consent.
* Pregnancy (suspected or known).

Risks of VCE VCE retention is the most dreaded adverse events. The risk may vary between 1.5 and 21%.

Allergic reactions may be possible due to the use of sticky electrodes on the skin.

Study duration 10 years from January 2016.

Confounders To date, not known.

Data management All results will remain confidential. Clinical data may become available at scientific meetings or in published articles, but patient anonymity will always be maintained

Statistics The incidence of neoplastic and preneoplastic lesions of the subjects included in the study will be estimated. The sample size was established on the basis of feasibility (10 subjects enrolled each year for each center in 10 years = 400 patients in total). The expected incidence of small bowel injury is approximately 5%. With 400 subjects it is possible to estimate the incidence with an accuracy of 2% estimated with a 95% confidence interval.

Descriptive statistical variables (mean, standard deviation, median, etc.) will be evaluated on the collected data.

Any relationships between these variables will be evaluated using inferential statistics (t-test, chi-squared, logistic regression analysis, multivariate analysis, etc.). Any relationship with a p-value less than 0.05 will be considered significant.

Ethics The investigators declare that the study will be conducted in accordance with the ethical principles deriving from the Declaration of Helsinki and the current legislation on Observational Studies.

Informed consent. All subjects will be informed of the purpose of the study, of the confidentiality of the personal data, and of the fact that this data may be subject to review, for study-related reasons, by authorized person other than the physician.

It will be emphasized that participation is entirely voluntary and that the patient can refuse further participation in the protocol at any time without affecting the patient's subsequent care. Informed consent will be obtained for all subjects included in the study prior to their inclusion in the present study, in accordance with national and local regulations.

ELIGIBILITY:
Inclusion Criteria:

* Pathogenic germline variant in one of the MMR genes (MLH1, MSH2/Epcam, MSH6, or PMS2).

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients unwilling or unable to provide informed consent
* Patients with prior small bowel surgery
* Patients with a contraindication to VCE

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Small bowel adenocarcinoma | 10 years
  Annual incidence
Small bowel adenoma | 10 years
  Annual incidence

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Scientific Institute, Gastroenterology and Gastrointestinal Endoscopy Unit, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lynch HT, Lynch PM, Lanspa SJ, Snyder CL, Lynch JF, Boland CR. Review of the Lynch syndrome: history, molecular genetics, screening, differential diagnosis, and medicolegal ramifications. Clin Genet. 2009 Jul;76(1):1-18. doi: 10.1111/j.1399-0004.2009.01230.x. PMID 19659756
- [Background] Koornstra JJ, Mourits MJ, Sijmons RH, Leliveld AM, Hollema H, Kleibeuker JH. Management of extracolonic tumours in patients with Lynch syndrome. Lancet Oncol. 2009 Apr;10(4):400-8. doi: 10.1016/S1470-2045(09)70041-5. PMID 19341971
- [Background] Koornstra JJ, Kleibeuker JH, Vasen HF. Small-bowel cancer in Lynch syndrome: is it time for surveillance? Lancet Oncol. 2008 Sep;9(9):901-5. doi: 10.1016/S1470-2045(08)70232-8. PMID 18760246
- [Background] ten Kate GL, Kleibeuker JH, Nagengast FM, Craanen M, Cats A, Menko FH, Vasen HF. Is surveillance of the small bowel indicated for Lynch syndrome families? Gut. 2007 Sep;56(9):1198-201. doi: 10.1136/gut.2006.118299. Epub 2007 Apr 4. PMID 17409122
- [Background] Rodriguez-Bigas MA, Vasen HF, Lynch HT, Watson P, Myrhoj T, Jarvinen HJ, Mecklin JP, Macrae F, St John DJ, Bertario L, Fidalgo P, Madlensky L, Rozen P. Characteristics of small bowel carcinoma in hereditary nonpolyposis colorectal carcinoma. International Collaborative Group on HNPCC. Cancer. 1998 Jul 15;83(2):240-4. doi: 10.1002/(sici)1097-0142(19980715)83:23.0.co;2-u. PMID 9669805
- [Background] Haanstra JF, Al-Toma A, Dekker E, Vanhoutvin SA, Nagengast FM, Mathus-Vliegen EM, van Leerdam ME, de Vos tot Nederveen Cappel WH, Sanduleanu S, Veenendaal RA, Cats A, Vasen HF, Kleibeuker JH, Koornstra JJ. Prevalence of small-bowel neoplasia in Lynch syndrome assessed by video capsule endoscopy. Gut. 2015 Oct;64(10):1578-83. doi: 10.1136/gutjnl-2014-307348. Epub 2014 Sep 10. PMID 25209657
- [Background] Saurin JC, Pilleul F, Soussan EB, Maniere T, D'Halluin PN, Gaudric M, Cellier C, Heresbach D, Gaudin JL; Capsule Commission of the French Society of Digestive Endoscopy (SFED). Small-bowel capsule endoscopy diagnoses early and advanced neoplasms in asymptomatic patients with Lynch syndrome. Endoscopy. 2010 Dec;42(12):1057-62. doi: 10.1055/s-0030-1255742. Epub 2010 Sep 6. PMID 20821360